CLINICAL TRIAL: NCT06933602
Title: The Impact of Progressive Relaxation Exercise Training on Hospital-Acquired Insomnia and Satisfaction Levels in COPD Patients
Brief Title: Progressive Relaxation for COPD: Effects on Insomnia and Satisfaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceylan Aksoy (Other)
Responsible Party: Sponsor-Investigator, Ceylan Aksoy, LECTURER, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-95531838-050.99-116055
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: COPD; Insomnia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Initiation and Maintenance Disorders | interventions — Relaxin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Implementation of Progressive Muscle Relaxation Training
  Interventions: Other: relaxin
- Control Group (No Intervention)

INTERVENTIONS:
Other: relaxin — Progressive Muscle Relaxation (PMR) exercises help alleviate symptoms in patients with COPD by reducing the effects of anxiety and stress, distracting attention from pain, and relieving muscle tension and spasms.
  These exercises are beneficial in managing:
  Tension headaches Back pain Tension and pain in jaw muscles Tension and pain around the eye muscles Muscle spasms Insomnia Stress-related muscle tension The required content of the exercises for relieving stress-related tension will be provided in a booklet. The booklet will be given to the patients following the training session.
  Arms: Intervention Group

SUMMARY:
In the life model based on the activities of living developed by nursing theorists Roper, Logan, and Tierney, sleep is identified as one of the twelve essential activities. Sleep is a fundamental need initiated by the circadian rhythm and sleep/wake homeostatic pressure, and it is followed by a period of wakefulness. Therefore, early identification of sleep disorders and the improvement of sleep and quality of life should be primary goals. As sleep quality improves, individuals feel better both physically and mentally; however, in individuals with Chronic Obstructive Pulmonary Disease (COPD), sleep problems tend to increase as symptoms worsen.

Non-pharmacological methods such as breathing exercises, reflexology, relaxation exercises, and physical exercises are commonly used to cope with symptoms in individuals with COPD. Among these, progressive muscle relaxation exercises (PMRE) have recently become an important component in the care of individuals with chronic illnesses, due to their benefits in reducing anxiety and stress, diverting attention from pain, and alleviating muscle tension and contractions.

Patient education, which is a component of the nurse's role as an educator, aims to help the patient prevent complications, gain self-sufficiency in daily life, cope with illnesses, adapt to the disease, and improve decision-making abilities. In addition to these numerous benefits, patient education also contributes to increased patient satisfaction. Progressive muscle relaxation training, by increasing body awareness-such as recognizing which muscles are located in which areas and how they react under stress-is considered an important educational tool that can enhance the patient's adaptation to the illness and assist in coping with symptoms.

The study will be conducted as a randomized controlled trial with a pretest-posttest experimental design. The sample will consist of a total of 70 patients-35 in the experimental group and 35 in the control group-who have been diagnosed with COPD at the Department of Chest Diseases in Van Yüzüncü Yıl University Dursun Odabaş Medical Center, meet the research criteria, and agree to participate in the study.

To ensure randomization, a dice-rolling method will be used. Each patient meeting the inclusion criteria will roll a die: if an odd number appears on the upper face, the patient will be assigned to the control group; if an even number, to the experimental group.

Both the experimental and control groups will be administered the Patient Information Form and the Insomnia Severity Index for Hospitalized Patients as pretests. In addition, the Patient Satisfaction with Education Scale will be applied as a posttest only to the experimental group.

While patients in the experimental group will be provided with an educational booklet and receive progressive muscle relaxation training, patients in the control group will receive routine nursing care and standard treatment without any additional training.

One week later, both groups will again be administered the Patient Information Form and the Insomnia Severity Index for Hospitalized Patients as posttests.

Data obtained from the study will be analyzed using the SPSS (Statistical Package for the Social Sciences) version 23.0 software.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with chronic obstructive pulmonary disease (COPD)

Exclusion Criteria:

* participants must not be under 18 years of age.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-22 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Hospital-Related Insomnia Scale: | 7 day
  The Hospital-Related Insomnia Scale was developed by Çiftçi, Yıldız, and Yıldız (2023) to assess patients' levels of insomnia caused by hospital-related factors. The scale consists of 18 items and five subdimensions: physical environmental factors (items 1-5), psychological factors (items 6-9), safety factors (items 10-12), socio-economic factors (items 13-15), and nutritional factors (items 16-18). The Cronbach's alpha reliability coefficients for the subdimensions were 0.842, 0.804, 0.786, 0.677, and 0.672 respectively, while the overall internal consistency of the scale was found to be 0.783. The scale is evaluated by calculating the average score of the items, with scores ranging from 1 to 5. Higher scores indicate greater levels of hospital-related insomnia associated with the corresponding factor.

CONTACTS AND LOCATIONS:
Locations (1):
- Ağrı İbrahim Çeçen University, Ağrı, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No